CLINICAL TRIAL: NCT01383707
Title: A Multi-center, Open-label Clinical Trial to Evaluate the Objective Response Rate of Bevacizumab in Combination With Modified FOLFOX-6 Followed by One Year of Maintenance With Bevacizumab Alone in Patients With Initially Not or Borderline Resectable Colorectal Liver Metastases (The CLMO-001 Trial)
Brief Title: A Study of Bevacizumab and Modified FOLFOX-6 (mFOLFOX-6) in Participants With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25625; 2011-001364-22 (EudraCT Number)
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Leucovorin; Oxaliplatin

ARMS (1):
- Bevacizumab + mFOLFOX-6 (Experimental): Participants will receive combination therapy of bevacizumab 5 mg/kg IV dose and mFOLFOX-6 (Levofolinic acid, 5-FU and oxaliplatin) on Day 1 of every 2 weeks' cycle for 5 cycles (Cycle 1-5), followed by 1 cycle (Cycle 6) of mFOLFOX6 alone (preoperative treatment phase). After 3 weeks of preoperative treatment phase, participants satisfying the surgical criteria for hepatic resectability will undergo a liver metastasectomy. Thereafter participants will receive combination therapy of mFOLFOX-6 + bevacizumab for another 6 cycles (Cycle 7-12); (post-operative treatment phase) followed by bevacizumab alone for 52 weeks (26 cycles) (maintenance therapy).
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Bevacizumab; Drug: Levofolinic acid; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-Fluorouracil (5-FU) — Participants will receive 5-FU 400 mg per meter-squared (mg/m^2) IV dose on Day 1 of each 2 weeks' cycle followed by 2400 mg/m^2, continuous infusion over 46 hours up to 12 cycles.
Drug: Bevacizumab — Participants will receive 5 mg/kg bevacizumab IV dose on Day 1 of each 2 weeks' cycle up to Cycle 5 and thereafter cycles 7 to 12; followed by maintenance therapy of 5 mg/kg IV every 2 weeks up to 52 weeks (26 cycles).
  Other Names: Avastin
Drug: Levofolinic acid — Participants will receive levofolinic acid 200 mg/m^2 IV infusion over 2 hours on Day 1 of each 2 weeks' cycle up to 12 cycles.
Drug: Oxaliplatin — Participants will receive oxaliplatin 85 mg/m^2 IV infusion over 2 hours on Day 1 of each 2 weeks' cycle up to 12 cycles.

SUMMARY:
The multicenter, open-label, single-arm, non-randomized, two-stage Simon's design, phase II study (The CLMO-001 Trial) will evaluate the efficacy and safety of bevacizumab in combination with mFOLFOX-6 (Levofolinic acid, 5-Fluorouracil [5-FU] and oxaliplatin) in participants with colorectal cancer and liver metastases. Participants will receive combination therapy of bevacizumab 5 milligrams per kilogram (mg/kg) intravenous (IV) dose and mFOLFOX-6 every 2 weeks during Cycles 1-5 and Cycles 7-12. Participants will receive mFOLFOX-6 alone (without bevacizumab) on Cycle 6. In between Cycle 6 and 7, participants will undergo liver surgery if operable. Thereafter participants will receive bevacizumab (5 mg/kg IV every 2 weeks) alone for 52 weeks (26 cycles) after the end of the post-operative phase (maintenance therapy). At the end of the preoperative treatment phase (Cycles 1-6), participants showing different alternative conditions admitted by the protocol will undergo different management (alternative study designs 1 to 3).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (male or female), greater than (>) 18 years of age
* Histologically confirmed adenocarcinoma of the colon or the rectum
* Primitive lesion is at a distance >12 centimeter (cm) from the anal margin for participants with primitive rectal tumor
* Measurable metastatic disease confined to the liver
* Eastern cooperative oncology group (ECOG) performance status 0-1
* No previous chemotherapy for metastatic disease or treatment with drugs targeting vascular endothelial growth factor receptor (VEGF) or epidermal growth factor receptor (EGFR)
* Adequate bone marrow, liver and renal function
* Urine analysis with proteinuria less than (<) 2+
* Use of at least one approved contraceptive method by participants with reproductive potential
* Written informed consent from the participants
* Surgical criteria for hepatic resection
* Adjuvant treatment (either only surgery on primitive tumor or surgery on primitive tumor + adjuvant chemotherapy) must have been concluded greater than or equal to (>/=) 6 months before enrollment

Exclusion Criteria:

* Presence of extrahepatic metastases
* Evidence of lumbo-aortic and celiac lymph nodes involvement
* Radiotherapy within 4 weeks before study start
* History of inflammatory bowel disease and/or acute/sub-acute bowel occlusion
* Presence of serious non-healing wound or ulcer
* Evidence of bleeding diathesis or coagulopathy
* Clinically significant cardiovascular disease
* Uncontrolled hypertension
* Current or recent ongoing treatment with anticoagulants
* Chronic, daily treatment with high-dose aspirin (>325 mg/day) or other medications known to predispose to gastrointestinal ulceration
* Treatment with any investigational drug within 30 days prior to enrollment
* Known allergy to Chinese hamster ovary cell proteins, or any of the components of the study medications
* Co-existing malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study. Interval between endoscopic biopsy or colorectal stenting and bevacizumab administration should be evaluated by oncologist/endoscopist
* Pregnant or lactating women
* Any other disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complication
* Participants with known Human immunodeficiency virus (HIV) infection
* Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection with concomitant cirrhosis or undergoing active treatment for the same
* Participants who are unable or unwilling to comply with the requirements of the protocol and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-08-12 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2016-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Italy (11):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica A, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - Azienda Ospedaliera Sant' Antonio Abate; Divisione di Oncologia, Gallarate, Lombardy
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima; Oncologia Medica, Catania, Sicily
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - Ospedali Riuniti Di Ancona; Oncology, Ancona, The Marches

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Modified FOLFOX-6 (mFOLFOX-6): Combination therapy of bevacizumab and mFOLFOX-6 (Levofolinic acid, 5-Fluorouracil [5-FU], oxaliplatin) on Day 1 of every 2 weeks' cycle for 5 cycles (Cycle 1-5), followed by 1 cycle (Cycle 6) of mFOLFOX6 alone (preoperative treatment phase). After 3 weeks of preoperative treatment phase, participants satisfying the surgical criteria for hepatic resectability will undergo a liver metastasectomy. Thereafter participants will receive combination therapy of mFOLFOX-6 + bevacizumab for another 6 cycles (Cycle 7-12); (post-operative treatment phase) followed by bevacizumab alone for 52 weeks (26 cycles) (maintenance therapy). 5-FU: 400 mg/meter-squared (mg/m^2) IV dose on Day 1 of each 2 weeks' cycle followed by 2400 mg/m^2, continuous infusion over 46 hours; Bevacizumab: 5 mg/kg IV on Day 1 of each 2 weeks' cycle; Levofolinic acid: 200 mg/m^2 IV infusion over 2 hours on Day 1 of each 2 weeks' cycle; Oxaliplatin: 85 mg/m^2 IV infusion over 2 hours on Day 1 of each 2 weeks' cycle
Period: Overall Study
Arm/Group | Bevacizumab + Modified FOLFOX-6 (mFOLFOX-6)
Started | 77
Completed | 5
Not Completed | 72
Not completed — Consent withdrawal | 6
Not completed — Death | 19
Not completed — Other | 8
Not completed — Sponsor's decision | 2
Not completed — Adverse Event | 14
Not completed — Progressive disease | 23

BASELINE CHARACTERISTICS:
Population: The intent-to-treat analysis set (ITT), which included all enrolled participants, who received at least one dose of any study medication.
Groups:
- Bevacizumab + mFOLFOX-6: Combination therapy of bevacizumab and mFOLFOX-6 (Levofolinic acid, 5-Fluorouracil [5-FU], oxaliplatin) on Day 1 of every 2 weeks' cycle for 5 cycles (Cycle 1-5), followed by 1 cycle (Cycle 6) of mFOLFOX6 alone (preoperative treatment phase). After 3 weeks of preoperative treatment phase, participants satisfying the surgical criteria for hepatic resectability will undergo a liver metastasectomy. Thereafter participants will receive combination therapy of mFOLFOX-6 + bevacizumab for another 6 cycles (Cycle 7-12); (post-operative treatment phase) followed by bevacizumab alone for 52 weeks (26 cycles) (maintenance therapy). 5-FU: 400 mg/meter-squared (mg/m^2) IV dose on Day 1 of each 2 weeks' cycle followed by 2400 mg/m^2, continuous infusion over 46 hours; Bevacizumab: 5 mg/kg IV on Day 1 of each 2 weeks' cycle; Levofolinic acid: 200 mg/m^2 IV infusion over 2 hours on Day 1 of each 2 weeks' cycle; Oxaliplatin: 85 mg/m^2 IV infusion over 2 hours on Day 1 of each 2 weeks' cycle
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in the Intent-to-treat (ITT) Analysis Set
Description: ORR was defined as the percentage of participants with shrinkage (partial response [PR]) or disappearance of cancer (complete response [CR]). Tumor response was evaluated according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). The same method of tumor measurement and assessment had to be used to characterize each lesion throughout the study. Tumor assessment consisted of computerized tomography (CT) scan (abdomen + pelvis + chest) or contrast-enhanced magnetic resonance imaging (CE-MRI) (abdomen + pelvis) + non CE-CT (chest) according to the choice of the center. CR, Disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 11 cycles of treatment (up to Week 22)
Population: The ITT set, which included all enrolled participants, who received at least one dose of any study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 77
percentage of participants | 54.5 [42.8 to 65.9]

2. Primary Outcome: Objective Response Rate (ORR) in the Per-protocol Analysis Set (PPAS)
Description: ORR was defined as the percentage of participants with shrinkage (PR) or disappearance of cancer (CR). Tumor response was evaluated according to the RECIST v1.1. The same method of tumor measurement and assessment had to be used to characterize each lesion throughout the study. Tumor assessment consisted of CT scan (abdomen + pelvis + chest) or CE-MRI (abdomen + pelvis) + non CE-CT (chest) according to the choice of the center. CR, Disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR.
Time Frame: Up to 11 cycles of treatment (up to Week 22)
Population: The PPAS included all subjects in the ITT set, who did not experience any major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 64
percentage of participants | 64.1 [51.1 to 75.7]

3. Secondary Outcome: Percentage of Participants Achieving No Residual Tumor (R0)/Surgical Margin With Microscopic Residual Tumor (R1) Liver Resection
Description: The percentage of participants achieving R0/R1 liver resection was defined as the percentage of participants achieving R0 surgery (no residual tumor) plus percentage of participants achieving R1 surgery (surgical margin with microscopic residual tumor).
Time Frame: End of study up to approximately 3 years
Population: The ITT set, which included all enrolled participants, who received at least one dose of any study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 77
percentage of participants | 29.9 [20.0 to 41.4]

4. Secondary Outcome: Disease-free Interval (DFI)
Description: DFI was defined as the time from the date of R0/R1 surgery to the date of disease relapse or death due to any cause. Participants who did not progress were considered censored at the date of the last assessment performed. For participants receiving two-stage resection, the date of R0/R1 surgery was the date of the second surgery. Participants, who did not receive surgery and participants without R0/R1 surgery were censored at Day 1. DFI was calculated as follows: DFI (months) = ([Date of R0/R1 surgery - Date of 1st relapse/Death] + 1)/30
Time Frame: End of study up to approximately 3 years
Population: The ITT set, which included all enrolled participants, who received at least one dose of any study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 77
months | 10.8 [5.7 to 15.7]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first study drug administration to the date of disease progression or death due to any cause, whichever came first. Progression was defined according to RECIST, v1.1 as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions. Participants, who did not progress were censored at the date of the last assessment performed. Participants who withdrew from the study without documented progression and for whom an electronic case report form (eCRF) existed as evidence that evaluations had been made, were censored at the date of the last tumor assessment when the participant was known to be progression-free. Participants without post-baseline tumor assessments, but known to be alive were censored at the time of first study drug administration. PFS was calculated: PFS (months) = ([Date of Event - Date of first study drug administration] + 1)/30.
Time Frame: End of study up to approximately 3 years
Population: The ITT set, which included all enrolled participants, who received at least one dose of any study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 77
months | 11.7 [10.3 to 14.3]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first study drug administration to the date of death due to any cause. Participants who were alive at the time of the analysis were censored at the last date the participant was known to be alive. OS was calculated as follows: OS (months) = ([Date of Death - first study drug administration] + 1)/30
Time Frame: End of study up to approximately 3 years
Population: The ITT set, which included all enrolled participants, who received at least one dose of any study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 77
months | NA [NA to NA] — The median overall survival time and its 95% confidence interval were not estimable because of the low number of events (less than 50%) and of the distribution of censored participants over time.

ADVERSE EVENTS:
Time Frame: End of study up to approximately 3 years.
Description: The safety analysis set (SAF) included all enrolled participants, who received at least one dose of any study medication. If there was any doubt whether a subject was treated or not, they were to be assumed treated for the purposes of analysis.
Arm/Group | Bevacizumab + mFOLFOX-6
Serious Adverse Events (participants affected / at risk) | 32/77
Other Adverse Events (participants affected / at risk) | 77/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + mFOLFOX-6 (N=77)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Biliary tract disorder (Hepatobiliary disorders) | 1
Biloma (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Subcutaneous abscess (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Biliary drainage (Surgical and medical procedures) | 1
Colectomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + mFOLFOX-6 (N=77)
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 17
Haemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 39
Stomatitis (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 32
Fatigue (General disorders) | 8
Mucosal inflammation (General disorders) | 9
Pyrexia (General disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 8
Neuropathy peripheral (Nervous system disorders) | 4
Neurotoxicity (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 44
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Erythema (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 30
Dyspepsia (Gastrointestinal disorders) | 4
White blood cell count decreased (Investigations) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 6
Proteinuria (Renal and urinary disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.